CLINICAL TRIAL: NCT02164487
Title: Evaluating the B1 Status in Eating Disorder Female Adolescent Patients
Brief Title: Thiamin (Vitamin B1) Levels in Eating Disorder Adolescent Patients
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, medical center research, Assaf-Harofeh Medical Center
Other Study IDs: 214/12
Record Dates: First submitted 2013-06-06; First posted 2014-06-16 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Eating Disorders
Keywords: B1 adolescents Eating disorders Thaimine
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- B1 blood levels

SUMMARY:
Vitamin B1 (Thiamine) is a water soluble essential nutrient; it is synthesized by a variety of plants and microorganisms. Since animals usually cannot synthesis it, humans must be supplied with exogenous vitamin B1 in the diet. The human storage of thiamine is small- about 30mg, an intake of 1-2 mg a day is needed to maintain this pool. Deficiency might occur when the vitamin is depleted from the diet in a short period. Vitamin B1 has a role in energy metabolism and main biosynthetic pathways. Low thiamine causes illnesses in the central and peripheral nervous systems as well as affecting the heart and gastrointestinal systems.

Deficiency may occur from malnutrition of different mechanisms such as alcoholism, lack in diet and recently secondary to anti-obesity surgery and few case reports described eating disorders as the reason for developing deficiency causing neuropathy, (1,2) and encephalopathy (3,4,5).

One of the presentations of thiamine deficiency is peripheral neuropathy mimicking Guillain-Barre syndrome, and administering the lacking vitamin improves the symptoms.

One study examined the prevalence of vitamin B1 deficiency in adult anorexia nervosa patients (6) by measurement of the activation of the enzyme erythrocyte transketolase following addition of thiamin pyrophosphate and comparing them to control of blood donors. This study found significant lower levels of vitamin B1 in the anorectic patient compared to the controls.

Rational of the study:

The investigators assume that these few cases described of overt neurologic impairment due to vitamin B1 deficiency because of distorted eating are just the "tip of the iceberg" and more eating disorders patients lack thiamine, that may have neuropsychiatric effect on the illness and identifying and treating the shortage may improve the symptoms of the disorder and maybe even the distorted thoughts that are fundamental in eating disorders.

DETAILED DESCRIPTION:
Methods:

In Assaf Harofe medical center over 50 adolescents (mainly girls) aged 10-18 years are treated annually for eating disorders by a multidisciplinary team. Their nutritional and medical condition is assessed also by blood analysis routinely. The investigators are planning to check thiamine status in eating disorders female patients in different stages of treatment, comparing them with age and sex matched controls that do not have eating disorders problems. The control group will be recruited from patient treated in the outpatient day hospital and have blood tested anyhow that don't suffer from eating, metabolic, nutritional or gastrointestinal disorders.

The researchers will look for correlation between different types of eating disorders, nutritional state, treatment progress and levels of vitamin B1.

Thiamin will be determined in whole blood using High-Performance Liquid Chromatography (HPLC) that is superior to the previous method as described above, determining thiamin diphosphate; the physiologically active form of vitamin B1 accurately.

Sample size: A previous study on thiamine concentration in 50 healthy French volunteers found a standard deviation (SD) of 15 nmol/l (7). 17 patients in each group were required in order to detect a 15 nmol/l difference in mean thiamine levels with a power of 80% and Alfa of 0.05. In order to overcome a possibly higher SD and to allow for subgroup analysis , we decided to recruit 30 patients for each group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls aged 12-18

Exclusion Criteria:

* Girls suffering from metabolic
* Nutritional or gastrointestinal disorders

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: adolescent girls with eating disordes aged 12-18
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
establishing B1 levels | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric devision Assaf harofeh MC, Zrifin, Israel